CLINICAL TRIAL: NCT01276509
Title: A Double-blind, Randomized, Placebo-controlled, Dose-ranging Study To Evaluate The Efficacy And Safety Of Pf-00547659 In Subjects With Crohn's Disease (Opera)
Brief Title: Study To Test Whether PF-00547659 Is Safe And Improves Disease Symptoms In Patients With Crohn's Disease
Acronym: OPERA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A7281006; 2010-023437-30 (EudraCT Number); OPERA (Other: Alias Study Number)
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Results first posted 2017-04-13 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease Safety Efficacy Pharmacokinetics Pharmacodynamics Crohn's Disease Activity Index (CDAI)
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo-SC Injection (Placebo Comparator): Placebo delivered SC, 3 doses separated by 4 weeks.
  Interventions: Drug: PF-00547659 SC injection
- Drug Dose level 1- SC injection (Experimental): Drug dose level 1 delivered SC, 3 doses separated by 4 weeks.
  Interventions: Drug: PF-00547659 SC injection
- Drug Dose level 2-SC injection (Experimental): Drug dose level 2 delievered SC, 3 doses separated by 4 weeks.
  Interventions: Drug: PF-00547659 SC injection
- Drug Dose level 3- SC injection (Experimental): Drug dose level 3 delivered SC, 3 doses separated by 4 weeks.
  Interventions: Drug: PF-00547659 SC injection

INTERVENTIONS:
Drug: PF-00547659 SC injection — Placebo delivered SC, 3 doses separated by 4 weeks
  Arms: Placebo-SC Injection
Drug: PF-00547659 SC injection — Drug dose level 1 delivered SC, 3 doses separated by 4 weeks
  Arms: Drug Dose level 1- SC injection
Drug: PF-00547659 SC injection — Drug dose level 2 delivered SC, 3 doses separated by 4 weeks
  Arms: Drug Dose level 2-SC injection
Drug: PF-00547659 SC injection — Drug dose level 3 delivered SC, 3 doses separated by 4 weeks
  Arms: Drug Dose level 3- SC injection

SUMMARY:
Adults with Crohn's disease that is clinically active despite conventional treatment will be eligible for this study. Patients may receive one of three doses of PF-00547659 (experimental drug) or placebo (inactive drug). Disease activity will be measured every two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have failed or are intolerant to anti-TNFs and/or immunosuppressants (AZA, 6-MP, and/or MTX).
* hsCRP greater than 3mg/L
* Ulcerations demonstrated by colonoscopy performed during screening or 8 weeks prior to screening

Exclusion Criteria:

* Pregnant or breast feeding
* Short bowel syndrome due to multiple small bowel resections
* Presence of a stoma

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2011-04-06 (Actual); Primary Completion 2014-02-07 (Actual); Study Completion 2015-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (137):
- United States (69):
  - Clopton Clinic, Jonesboro, Arkansas
  - Gastroenterology Specialists of Arkansas, Jonesboro, Arkansas
  - Little Rock Diagnostic Clinic, P.A., Little Rock, Arkansas
  - UCSD Medical Center-Thornton Hospital, La Jolla, California
  - Community Clinical Trials, Orange, California
  - Gastro Diagnostics, Orange, California
  - Inland Gastroenterology Medical Associates, Inc., Redlands, California
  - BioMark Research Inc., Whittier, California
  - Clinical Research of the Rockies, Lafayette, Colorado
  - Rocky Mountain Gastroenterology Associates, Thornton, Colorado
  - Connecticut Clinical Research Foundation, Bristol, Connecticut
  - Shands Endoscopy Center, Gainesville, Florida
  - Shands Hospital at the University of Florida, Gainesville, Florida
  - Shands Medical Plaza, Gainesville, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Florida Center for Gastroenterology, Largo, Florida
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - University of Miami Hospital and Clinic, Miami, Florida
  - University of Miami Hospital, Miami, Florida
  - University of Miami, Miami, Florida
  - Cirtus Ambulartory Surgery Center, Orlando, Florida
  - Internal Medicine Specialists, Orlando, Florida
  - Heartland Medical Research (Administrative Only), Clive, Iowa
  - Iowa Digestive Disease Center, Clive, Iowa
  - Iowa Endoscopy Center (Colonoscopy Only), Clive, Iowa
  - Metropolitan Gastroenterology Group, PC - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - University of Massachusetts Worcester, Worcester, Massachusetts
  - Center for Digestive Health, Troy, Michigan
  - Surgical Centers of Michigan, Troy, Michigan
  - Minneapolis Heart Institute, West Health Campus, Minneapolis, Minnesota
  - Noran Neurology Clinic, Minneapolis, Minnesota
  - Consulting Radiology (Xray testing only), Plymouth, Minnesota
  - Minnesota Gastroenterology, P.A., Plymouth, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Surgery Center of Columbia, Columbia, Missouri
  - Audrain Medical Center, Mexico, Missouri
  - Center for Digestive and Liver Diseases, Inc., Mexico, Missouri
  - Barnes-Jewish Hospital - Investigational Drug Services, St Louis, Missouri
  - Center for Advanced Medicine, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Albany Medical College, Albany, New York
  - Life Medi-Research And Management, Brooklyn, New York
  - New York Hospital Queens, Flushing, New York
  - Long Island Clinical Research Associates, LLP, Great Neck, New York
  - Nassau Gastroenterology Associates Office Based Surgery, Great Neck, New York
  - Nassau Gastroenterology Associates, P.C., Great Neck, New York
  - North Shore Primary Care, P.C., Great Neck, New York
  - Beth Israel Medical Center - Phillip Ambulatory Care Center, New York, New York
  - East side Endoscopy, LLC (for colonscopy testing only), New York, New York
  - Lenox Hill Endoscopy Center, New York, New York
  - Premier Medical Group of the Hudson Valley, Poughkeepsie, New York
  - CTRC Hospital - UNC Memorial Hospital, Chapel Hill, North Carolina
  - North Carolina Memorial Hospital Endoscopy Center, Chapel Hill, North Carolina
  - UNC Hospitals Department of Pharmacy, Chapel Hill, North Carolina
  - UNC Hospitals Endoscopy, Chapel Hill, North Carolina
  - Hillsborough Campus, Hillsborough, North Carolina
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - The Offices of Dr. Vincent Armenio, M.D., East Providence, Rhode Island
  - Pharma Resource, East Providence, Rhode Island
  - Bayside Endoscopy Center, Providence, Rhode Island
  - Nashville Medical Research Institute, Nashville, Tennessee
  - Pasadena Gastroenterology Associates, P.A. dba Digestive Health Center, Pasadena, Texas
  - University of Utah HSC, Salt Lake City, Utah
  - Charlottesville Gastroenterology Associates, Charlottesville, Virginia
  - Charlottesville Medical Research, Charlottesville, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Allegiance Research Specialists, Wauwatosa, Wisconsin
  - GI Associates, Wauwatosa, Wisconsin
- AKH Wien Universitaetsklinik fuer Innere Medizin III, Vienna, Austria
- Belgium (4):
  - UZ Gasthuisberg, Leuven
  - Centre Hospitalier Universitaire de Liege, Liège
  - Centre Hospitalier Universitaire de Liège - Labo Biologie Clinique, Liège
  - Centre Hospitalier de Mouscron, Mouscron
- Bulgaria (2):
  - 4-MHAT, Sofia
  - MBAL Sofiamed OOD,Otdelenie po gastroenterologia, Sofia
- Canada (4):
  - Vancouver Coastal Health - Vancouver General Hospital, Vancouver, British Columbia
  - Vancouver Coastal Health - Vancouver Hospital, Vancouver, British Columbia
  - Oshawa Clinic, Oshawa, Ontario
  - Toronto Digestive Disease Associates Inc., Vaughan, Ontario
- France (8):
  - CHU Amiens Hopital Nord Service d'Hepato-Gastroenterologie, Amiens
  - Hopital Saint-Andre, Bordeaux
  - Hopital Beaujon- Essais cliniques, Clichy
  - Hopital de l'Archet 2 - CHU de Nice, Nice
  - Hopital Cochin-Essais Cliniques, Paris
  - Hopital Charles Nicolle, Rouen
  - Hopital Nord, Saint-Priest-en-Jarez
  - Hopital Rangueil, Toulouse
- Germany (8):
  - Charite - Campus Berlin Mitte Medizinische Klinik, Berlin
  - Krankenhaus Martha-Maria Halle-Doelau gGmbH, Halle
  - Universitaetsklinikum Schleswig-Holstein, Kiel
  - Universitaetsfrauenklinikum Schleswig-Holstein Medizinische Klinik I, Gastroenterologie/Hepatologie, Lübeck
  - Gastroenterologische Gemeinschaftspraxis Minden, Minden
  - Universitaetsklinikum Regensburg, Regensburg
  - Robert-Bosch-Krankenhaus, Stuttgart
  - Universitaetklinikum Ulm, Ulm
- Japan (7):
  - National Hospital Organization Hirosaki National Hospital, Hirosaki, Aomori
  - National Hospital Organization Takasaki General Medical Center, Takasaki, Gunma
  - Jikei University Hospital, Minato-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Aichi Medical University Hospital, Aichi
  - Chiba University Hospital, Chiba
  - Yokohama City University Medical Center, Kanagawa
- Netherlands (3):
  - Academic Medical Center, Amsterdam, North Holland
  - University Medical Center Groningen (UMCG), Groningen, Provincie Groningen
  - Maastricht University Medical Center, Maastricht
- Norway (3):
  - Asker And Baerum Hospital, Gjettum
  - Oslo Universitetssykehus, Oslo
  - Lovisenberg Diakonale Sykehus, Oslo
- Poland (4):
  - Szpital Uniwersytecki nr 2 im dr. Jana Bizieta w Bydgoszczy Centrum Endoskopii Zabiegowej, Bydgoszcz
  - Centrum Medyczne-Szpital Swietej Rodziny Sp. z o.o., Lodz
  - Centralny Szpital Kliniczny Ministerstwa Spraw Wewnetrznych w Warszawie, Warsaw
  - Lexmedica, Wroclaw
- Serbia (4):
  - Military Medical Academy, Belgrade
  - Clinical Hospital Centre Bezanijska Kosa, Belgrade
  - Clinical Center Nis Clinic for Gastroenterology and Hepatology, Niš
  - Clinical Hospital Center Zemun, Zemun
- Slovakia (4):
  - Gastroentero-Hepatologicke centrum THALION, LAMA MEDICAL CARE s.r.o., Bratislava
  - Medak s.r.o., Bratislava
  - Gastroenterologicke a hepatologicke centrum Nitra, KM Management spol. s r.o., Nitra
  - Synergy group, a.s., Nové Mesto nad Váhom
- South Africa (3):
  - Wits Clinical Research, Johannesburg, Gauteng
  - Parklands Medical Centre, Durban, KwaZulu-Natal
  - Kingsbury Hospital, Cape Town, Western Cape
- South Korea (7):
  - Pusan National University Hospital, Busan
  - Yeungnam University Hospital, Daegu
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Yonsei University College of Medicine, Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
- Spain (6):
  - Hospital Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitari Bellvitge, Barcelona
  - Hospital Universitario de La Princesa, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Corporacio Sanitaria Parc Tauli de Sabadell, Sabadell

REFERENCES:
- [Derived] Saruta M, Park DI, Kim YH, Yang SK, Jang BI, Cheon JH, Im JP, Kanai T, Katsuno T, Ishiguro Y, Nagaoka M, Isogawa N, Li Y, Banerjee A, Ahmad A, Hassan-Zahraee M, Clare R, Gorelick KJ, Cataldi F, Watanabe M, Hibi T. Anti-MAdCAM-1 antibody (PF-00547659) for active refractory Crohn's disease in Japanese and Korean patients: the OPERA study. Intest Res. 2020 Jan;18(1):45-55. doi: 10.5217/ir.2019.00039. Epub 2020 Jan 30. PMID 32013314
- [Derived] Sandborn WJ, Lee SD, Tarabar D, Louis E, Klopocka M, Klaus J, Reinisch W, Hebuterne X, Park DI, Schreiber S, Nayak S, Ahmad A, Banerjee A, Brown LS, Cataldi F, Gorelick KJ, Cheng JB, Hassan-Zahraee M, Clare R, D'Haens GR. Phase II evaluation of anti-MAdCAM antibody PF-00547659 in the treatment of Crohn's disease: report of the OPERA study. Gut. 2018 Oct;67(10):1824-1835. doi: 10.1136/gutjnl-2016-313457. Epub 2017 Oct 5. PMID 28982740
- [Derived] Hassan-Zahraee M, Banerjee A, Cheng JB, Zhang W, Ahmad A, Page K, von Schack D, Zhang B, Martin SW, Nayak S, Reddy P, Xi L, Neubert H, Fernandez Ocana M, Gorelick K, Clare R, Vincent M, Cataldi F, Hung K. Anti-MAdCAM Antibody Increases ss7+ T Cells and CCR9 Gene Expression in the Peripheral Blood of Patients With Crohn's Disease. J Crohns Colitis. 2018 Jan 5;12(1):77-86. doi: 10.1093/ecco-jcc/jjx121. PMID 28961803
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7281006&StudyName=Study%20To%20Test%20Whether%20PF-00547659%20Is%20Safe%20And%20Improves%20Disease%20Symptoms%20In%20Patients%20With%20Crohn%27s%20Disease

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In total, 265 participants were randomized and 262 entered the study and received study treatment.
Groups:
- PF-00547659 22.5 mg: PF-00547659 22.5 mg delivered subcutaneously (SC), 3 doses separated by 4 weeks.
- PF-00547659 75 mg: PF-00547659 75 mg delivered SC, 3 doses separated by 4 weeks
- PF-00547659 225 mg: PF-00547659 225 mg delivered SC, 3 doses separated by 4 weeks
- Placebo: Placebo delivered SC, 3 doses separated by 4 weeks.
Period: Overall Study
Arm/Group | PF-00547659 22.5 mg | PF-00547659 75 mg | PF-00547659 225 mg | Placebo
Started | 66 | 65 | 68 | 63
Completed | 53 | 53 | 63 | 58
Not Completed | 13 | 12 | 5 | 5
Not completed — Adverse Event | 9 | 8 | 4 | 3
Not completed — Lack of Efficacy | 2 | 1 | 1 | 2
Not completed — Pregnancy | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 0
Not completed — Other | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-00547659 22.5 mg | PF-00547659 75 mg | PF-00547659 225 mg | Placebo | Total
Number analyzed (Participants) | 66 | 65 | 68 | 63 | 262
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (13.0) | 34.4 (10.7) | 35.9 (11.0) | 34.4 (11.1) | 35.5 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 35 | 43 | 30 | 156
  Male | 18 | 30 | 25 | 33 | 106

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Crohn's Disease Activity Index (CDAI) 70 Response Rate
Description: Crohn's Disease Activity Index (CDAI) is a number which consists of information collected from a 7-day diary from the participants regarding symptoms. Remission is considered a score of 150 or less. Active disease is considered 200 or greater. A response to therapy is considered a decline in CDAI score of 70-points from baseline. CDAI response rate at week 8 and week 12 was measured between the investigational product group and the placebo group.
Time Frame: Week 8 and week 12
Population: The full analysis set included all randomized participants who received at least one dose of study medication.
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-00547659 22.5 mg | PF-00547659 75 mg | PF-00547659 225 mg | Placebo
Number analyzed (Participants) | 66 | 65 | 68 | 63
Percentage of Participants
  Week 8 (n =50, 55, 62, 56) | 52.7 | 60.1 | 62.7 | 47.7
  Week 12 (n = 51, 49, 61, 54) | 62.0 | 64.7 | 57.5 | 58.6
Statistical Analysis 1: Comparison: PF-00547659 22.5 mg vs Placebo; Difference from placebo at Week 8; Test type: Superiority or Other; p = 0.3393, Mixed Models Analysis; Difference in Percentage = 0.050, 90% CI 2-sided [-0.149 to 0.249], Standard Error of Mean 0.121
Statistical Analysis 2: Comparison: PF-00547659 75 mg vs Placebo; Difference from placebo at Week 8; Test type: Superiority or Other; p = 0.1433, Mixed Models Analysis; Difference in Percentage = 0.124, 90% CI 2-sided [-0.068 to 0.316], Standard Error of Mean 0.117
Statistical Analysis 3: Comparison: PF-00547659 225 mg vs Placebo; Difference from placebo at Week 8; Test type: Superiority or Other; p = 0.0922, Mixed Models Analysis; Difference in Percentage = 0.150, 90% CI 2-sided [-0.036 to 0.335], Standard Error of Mean 0.113
Statistical Analysis 4: Comparison: PF-00547659 22.5 mg vs Placebo; Difference from placebo at Week 12; Test type: Superiority or Other; p = 0.3864, Mixed Models Analysis; Difference in Percentage = 0.034, 90% CI 2-sided [-0.158 to 0.225], Standard Error of Mean 0.117
Statistical Analysis 5: Comparison: PF-00547659 75 mg vs Placebo; Difference from placebo at Week 12; Test type: Superiority or Other; p = 0.3005, Mixed Models Analysis; Difference in Percentage = 0.061, 90% CI 2-sided [-0.131 to 0.253], Standard Error of Mean 0.117
Statistical Analysis 6: Comparison: PF-00547659 225 mg vs Placebo; Difference from placebo at Week 12; Test type: Superiority or Other; p = 0.5385, Mixed Models Analysis; Difference in Percentage = -0.011, 90% CI 2-sided [-0.198 to 0.176], Standard Error of Mean 0.114

2. Secondary Outcome: Safety and Tolerability of PF-00547659 Dose Levels Versus Placebo
Description: Number of participants with adverse events (AEs), withdrawals due to AEs and Serious AEs (SAEs) were reported.
Time Frame: Week 0-12
Population: The safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: Number of participants
Arm/Group | PF-00547659 22.5 mg | PF-00547659 75 mg | PF-00547659 225 mg | Placebo
Number analyzed (Participants) | 66 | 65 | 68 | 63
Number of participants
  Participants with AEs (all causalities) | 57 | 51 | 54 | 54
  Participants with AEs (treatment related) | 20 | 24 | 29 | 22
  Withdrawal due to AEs (all causalities) | 9 | 8 | 4 | 3
  Withdrawal due to AEs (treatment related) | 5 | 2 | 0 | 1
  Participants with SAEs (all causalities) | 11 | 9 | 11 | 5
  Participants with SAEs (treatment related) | 4 | 4 | 2 | 2

3. Secondary Outcome: Number of Adverse Events (AEs) - PF-00547659 Dose Levels Versus Placebo
Description: Number of adverse events (all causalities and treatment related) was reported between the investigational product groups and the placebo group.
Time Frame: Week 0-12
Population: The safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: events
Arm/Group | PF-00547659 22.5 mg | PF-00547659 75 mg | PF-00547659 225 mg | Placebo
Number analyzed (Participants) | 66 | 65 | 68 | 63
events
  Number of AEs (all causalities) | 175 | 192 | 192 | 141
  Number of AEs (treatment related) | 40 | 55 | 64 | 40

4. Secondary Outcome: Percentage of Participants With a Crohn's Disease Activity Index (CDAI) Remission
Description: Percentage of participants with a CDAI remission (defined as a CDAI reduction to <150 points).
Time Frame: Weeks 8 and week 12
Population: The full analysis set included all randomized participants who received at least one dose of study medication.
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-00547659 22.5 mg | PF-00547659 75 mg | PF-00547659 225 mg | Placebo
Number analyzed (Participants) | 66 | 65 | 68 | 63
Percentage of Participants
  Week 8 (n = 50, 56, 62, 57) | 29.1 | 23.8 | 26.9 | 16.7
  Week 12 (n= 51, 49, 61, 55) | 26.8 | 28.5 | 29.6 | 23.0
Statistical Analysis 1: Comparison: PF-00547659 22.5 mg vs Placebo; Difference from placebo at week 8; Test type: Superiority or Other; p = 0.1234, Mixed Models Analysis; Difference in Percentage = 0.124, 90% CI 2-sided [-0.052 to 0.299], Standard Error of Mean 0.107
Statistical Analysis 2: Comparison: PF-00547659 75 mg vs Placebo; Difference from placebo at week 8; Test type: Superiority or Other; p = 0.2378, Mixed Models Analysis; Difference in Percentage = 0.071, 90% CI 2-sided [-0.092 to 0.234], Standard Error of Mean 0.099
Statistical Analysis 3: Comparison: PF-00547659 225 mg vs Placebo; Difference from placebo at week 8; Test type: Superiority or Other; p = 0.1529, Mixed Models Analysis; Difference in Percentage = 0.102, 90% CI 2-sided [-0.062 to 0.266], Standard Error of Mean 0.100
Statistical Analysis 4: Comparison: PF-00547659 22.5 mg vs Placebo; Difference from placebo at week 12; Test type: Superiority or Other; p = 0.3661, Mixed Models Analysis; Difference in Percentage = 0.038, 90% CI 2-sided [-0.146 to 0.222], Standard Error of Mean 0.112
Statistical Analysis 5: Comparison: PF-00547659 75 mg vs Placebo; Difference from placebo at week 12; Test type: Superiority or Other; p = 0.3169, Mixed Models Analysis; Difference in Percentage = 0.055, 90% CI 2-sided [-0.136 to 0.246], Standard Error of Mean 0.116
Statistical Analysis 6: Comparison: PF-00547659 225 mg vs Placebo; Difference from placebo at week 12; Test type: Superiority or Other; p = 0.2755, Mixed Models Analysis; Difference in Percentage = 0.066, 90% CI 2-sided [-0.116 to 0.248], Standard Error of Mean 0.111

5. Secondary Outcome: Crohn's Disease Activity Index (CDAI)-70 Response Rates Over Time
Description: Percentage of participants with Crohn's Disease Activity Index (CDAI)-70 response were reported.
Time Frame: Week 2, 4, 6, 8, 10 and 12
Population: The full analysis set included all randomized participants who received at least one dose of study medication.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | PF-00547659 22.5 mg | PF-00547659 75 mg | PF-00547659 225 mg | Placebo
Number analyzed (Participants) | 66 | 65 | 68 | 63
Percentage of Participants
  Week 2 (n = 64, 60, 63, 60) | 35.1 [22.8 to 49.6] | 22.4 [12.9 to 36.0] | 33.8 [21.6 to 48.5] | 35.5 [22.9 to 50.5]
  Week 4 (n = 58, 60, 65, 58) | 38.0 [24.9 to 53.2] | 39.5 [26.3 to 54.4] | 36.2 [23.7 to 51.0] | 38.3 [25.1 to 53.5]
  Week 6 (n =56, 54, 64, 58) | 45.3 [31.1 to 60.3] | 53.4 [38.2 to 67.9] | 47.5 [33.3 to 62.1] | 48.0 [33.5 to 62.9]
  Week 8 (n =50, 55, 62, 56) | 52.7 [37.2 to 67.7] | 60.1 [44.9 to 73.6] | 62.7 [47.9 to 75.4] | 47.7 [33.1 to 62.7]
  Week 10 (n =50, 48, 60, 52) | 67.4 [52.0 to 79.7] | 58.2 [42.3 to 72.6] | 61.6 [46.8 to 74.6] | 53.0 [37.6 to 67.8]
  Week 12 (n = 51, 49, 61, 54) | 62.0 [46.5 to 75.3] | 64.7 [48.9 to 77.8] | 57.5 [42.6 to 71.2] | 58.6 [43.3 to 72.4]

6. Secondary Outcome: Crohn's Disease Activity Index (CDAI) -100 Response Rates Over Timer
Description: Percentage of participants with Crohn's Disease Activity Index (CDAI)-100 response were reported.
Time Frame: Week 2, 4, 6, 8, 10 and 12
Population: The full analysis set included all randomized participants who received at least one dose of study medication.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | PF-00547659 22.5 mg | PF-00547659 75 mg | PF-00547659 225 mg | Placebo
Number analyzed (Participants) | 66 | 65 | 68 | 63
Percentage of Participants
  Week 2 (n = 64, 60, 63, 60) | 19.3 [10.6 to 32.6] | 18.4 [9.9 to 31.7] | 20.0 [11.0 to 33.6] | 18.5 [9.9 to 31.9]
  Week 4 (n = 58, 60 ,65, 58) | 29.2 [17.5 to 44.6] | 32.3 [20.0 to 47.5] | 28.2 [17.0 to 43.0] | 29.5 [17.7 to 44.9]
  Week 6 (n =56, 54, 64, 58) | 40.6 [26.6 to 56.4] | 42.6 [28.2 to 58.5] | 40.4 [26.8 to 55.8] | 39.3 [25.5 to 55.0]
  Week 8 (n = 50, 55, 62, 56) | 50.5 [34.8 to 66.2] | 48.3 [33.3 to 63.7] | 57.0 [41.8 to 71.0] | 41.4 [27.2 to 57.3]
  Week 10 (n = 50, 48, 62, 52) | 53.2 [37.3 to 68.5] | 47.4 [31.8 to 63.5] | 50.9 [35.9 to 65.7] | 43.6 [28.7 to 59.7]
  Week 12 (n = 51, 49, 61, 54) | 56.0 [40.1 to 70.7] | 47.7 [32.2 to 63.7] | 53.8 [38.7 to 68.4] | 44.4 [29.6 to 60.2]

7. Secondary Outcome: Immunogenicity Assessment of Anti-drug Antibodies (ADAs)
Description: Confirmed cumulative incidence of anti-drug antibodies development to PF-00547659
Time Frame: Day 1, Week 4, Week 8, Week 12, Week 20, Week 28, Week 36
Population: The safety analysis set included all participants who receive at least 1 dose of PF-00547659. Participants in placebo arm were not included in this analysis.
Measure: Number; unit: events
Arm/Group | PF-00547659 22.5 mg | PF-00547659 75 mg | PF-00547659 225 mg
Number analyzed (Participants) | 66 | 65 | 68
events
  Day 1 (n =46, 52, 53) | 3 | 5 | 1
  Week 4 (n = 55, 52, 55) | 2 | 4 | 2
  Week 8 (n = 44, 47, 56) | 1 | 1 | 1
  Week 12 (n = 47, 51, 51) | 3 | 5 | 1
  Week 20 (n = 4, 3, 1) | 0 | 0 | 0
  Week 28 (n = 8, 1, 1) | 1 | 0 | 0
  Week 36 (n = 6, 2, 1) | 0 | 0 | 0

8. Secondary Outcome: The Pharmacokinetics (PK) of Total PF-00547659 - Area Under the Concentration Time Profile From Time Zero Extrapolated to Infinite Time (AUCinf)
Description: The Pharmacokinetics (PK) of total PF-00547659 was characterized using a population PK approach. PK parameters including but not limited to area under the concentration-time profile (AUC), clearance (CL) and half life were estimated using data pooled from both typical and additional PK groups. AUCinf is area under the concentration time profile from time zero extrapolated to infinite time.
Time Frame: Day 1, 14, 28, 42, 56, 70, 84, 112, 140, 168, 196, 224 and 252
Population: All participants who received at least 1 dose of investigational product and had data for at least 1 PK concentration were included in the PK concentration analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg•hr/mL
Arm/Group | PF-00547659 22.5 mg | PF-00547659 75 mg | PF-00547659 225 mg
Number analyzed (Participants) | 6 | 8 | 6
µg•hr/mL | 615300 (63) | 4464000 (28) | 13760000 (49)

9. Secondary Outcome: The Pharmacokinetics (PK) of Total PF-00547659 - Area Under the Concentration Time Profile From Time Zero to Time Tau (AUCtau)
Description: The Pharmacokinetics (PK) of total PF-00547659 was characterized using a population PK approach. PK parameters including but not limited to AUC, CL and half life were estimated using data pooled from both typical and additional PK groups. AUCtau is area under the concentration time profile from time zero to time tau, the dosing interval, where tau = 672 hours (4 weeks)
Time Frame: Day 1, 14, and 28
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg•hr/mL
Arm/Group | PF-00547659 22.5 mg | PF-00547659 75 mg | PF-00547659 225 mg
Number analyzed (Participants) | 7 | 10 | 12
µg•hr/mL | 549500 (53) | 4214000 (31) | 10850000 (45)

10. Secondary Outcome: The Pharmacokinetics (PK) of Total PF-00547659 - Maximum Observed Concentration (Cmax)
Description: The Pharmacokinetics (PK) of total PF-00547659 was characterized using a population PK approach. PK parameters including but not limited to AUC, CL and half life were estimated using data pooled from both typical and additional PK groups. Cmax is maximum observed concentration.
Time Frame: Day 1, 14, 28, 42, 56, 70, 84, 112, 140, 168, 196, 224 and 252
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | PF-00547659 22.5 mg | PF-00547659 75 mg | PF-00547659 225 mg
Number analyzed (Participants) | 7 | 10 | 13
µg/mL | 1756 (45) | 10800 (22) | 24100 (47)

11. Secondary Outcome: The Pharmacokinetics (PK) of Total PF-00547659 - Time for Cmax (Tmax)
Description: The Pharmacokinetics (PK) of total PF-00547659 was characterized using a population PK approach. PK parameters including but not limited to AUC, CL and half life were estimated using data pooled from both typical and additional PK groups. Tmax is time for Cmax.
Time Frame: Day 1, 14, 28, 42, 56, 70, 84, 112, 140, 168, 196, 224 and 252
Population: as for outcome 8
Measure: Median (Full Range); unit: Hours
Arm/Group | PF-00547659 22.5 mg | PF-00547659 75 mg | PF-00547659 225 mg
Number analyzed (Participants) | 7 | 10 | 13
Hours | 140 (45) [43.9 to 333] | 143 (22) [44.9 to 171] | 165 (47) [51.7 to 214]

12. Secondary Outcome: The Pharmacokinetics (PK) of Total PF-00547659 - Terminal Half Life (Thalf)
Description: The Pharmacokinetics (PK) of total PF-00547659 was characterized using a population PK approach. PK parameters including but not limited to AUC, CL and half life were estimated using data pooled from both typical and additional PK groups. Thalf is terminal half life.
Time Frame: Day 1, 14, 28, 42, 56, 70, 84, 112, 140, 168, 196, 224 and 252
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Day
Arm/Group | PF-00547659 22.5 mg | PF-00547659 75 mg | PF-00547659 225 mg
Number analyzed (Participants) | 6 | 8 | 6
Day | 4.977 (2.8435) | 8.770 (2.3571) | 12.22 (3.8306)

13. Secondary Outcome: The Pharmacokinetics (PK) of Total PF-00547659 - Apparent Clearance (CL/F)
Description: The Pharmacokinetics (PK) of total PF-00547659 was characterized using a population PK approach. PK parameters including but not limited to AUC, CL and half life were estimated using data pooled from both typical and additional PK groups. CL/F is apparent clearance.
Time Frame: Day 1, 14, 28, 42, 56, 70, 84, 112, 140, 168, 196, 224 and 252
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hr
Arm/Group | PF-00547659 22.5 mg | PF-00547659 75 mg | PF-00547659 225 mg
Number analyzed (Participants) | 6 | 8 | 6
mL/hr | 36.54 (63) | 16.79 (28) | 16.38 (49)

ADVERSE EVENTS:
Arm/Group | PF-00547659 22.5 mg | PF-00547659 75 mg | PF-00547659 225 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 12/66 | 11/65 | 11/68 | 6/63
Other Adverse Events (participants affected / at risk) | 36/66 | 32/65 | 42/68 | 35/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-00547659 22.5 mg (N=66) | PF-00547659 75 mg (N=65) | PF-00547659 225 mg (N=68) | Placebo (N=63)
Abdominal adhesions (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 5 | 6 | 4 | 4
Fistula of small intestine (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Rectal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Subileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 1 | 1
Appendicitis (Infections and infestations) | 2 | 0 | 0 | 0
Liver abscess (Infections and infestations) | 1 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1 | 0
Rectal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-00547659 22.5 mg (N=66) | PF-00547659 75 mg (N=65) | PF-00547659 225 mg (N=68) | Placebo (N=63)
Abdominal pain (Gastrointestinal disorders) | 7 | 1 | 4 | 3
Crohn's disease (Gastrointestinal disorders) | 5 | 7 | 1 | 5
Diarrhoea (Gastrointestinal disorders) | 1 | 4 | 1 | 1
Nausea (Gastrointestinal disorders) | 7 | 4 | 5 | 7
Proctalgia (Gastrointestinal disorders) | 1 | 4 | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 3 | 3 | 4
Fatigue (General disorders) | 5 | 4 | 2 | 3
Injection site erythema (General disorders) | 1 | 4 | 2 | 3
Oedema peripheral (General disorders) | 0 | 1 | 5 | 0
Pyrexia (General disorders) | 5 | 6 | 8 | 7
Influenza (Infections and infestations) | 4 | 2 | 1 | 1
Nasopharyngitis (Infections and infestations) | 3 | 4 | 5 | 5
Urinary tract infection (Infections and infestations) | 2 | 1 | 3 | 5
Vulvovaginal mycotic infection (Infections and infestations) | 3 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 6 | 5 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4 | 2
Headache (Nervous system disorders) | 6 | 3 | 8 | 6
Erythema (Skin and subcutaneous tissue disorders) | 3 | 2 | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other